CLINICAL TRIAL: NCT02648776
Title: Risk and Benefit Assessment of Hypnotic Agents for Sleep Disorders Among Elderly; A Prospective Cohort Study at a Taiwanese Academic Medical Center
Brief Title: Risk and Benefit Assessment of Hypnotic Agents for Sleep Disorders Among Elderly
Acronym: RABA-HASDE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: China Medical University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Hsiang-Wen Lin, Associate Professor, China Medical University Hospital
Other Study IDs: DMR101-IRB1-083
Record Dates: First submitted 2015-03-24; First posted 2016-01-07 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Sleep Disorders
Keywords: hypnotic agents; sleep disorders; elderly
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A single set of blood and urine samples taken in cohorts taking sedative-hypnotic medications, used to evaluate pharmacokinetic and pharmcogenetic parameters.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- Estazolam: Exposure to sedative-hypnotic drugs; Patients who have taken estazolam for at least one week before the first date of enrollment
  Interventions: Drug: Exposure to sedative-hypnotic drugs
- Lorazepam: Exposure to sedative-hypnotic drugs; Patients who have taken lorazepam for at least one week before the first date of enrollment
  Interventions: Drug: Exposure to sedative-hypnotic drugs
- Diazepam: Exposure to sedative-hypnotic drugs; Patients who have taken Diazepam for at least one week before the first date of enrollment
  Interventions: Drug: Exposure to sedative-hypnotic drugs
- Alprazolam: Exposure to sedative-hypnotic drugs; Patients who have taken Alprazolam for at least one week before the first date of enrollment
  Interventions: Drug: Exposure to sedative-hypnotic drugs
- Flunitrazepam: Exposure to sedative-hypnotic drugs; Patients who have taken Flunitrazepam for at least one week before the first date of enrollment
  Interventions: Drug: Exposure to sedative-hypnotic drugs
- Zolpidem: Exposure to sedative-hypnotic drugs; Patients who have taken Zolpidem for at least one week before the first date of enrollment
  Interventions: Drug: Exposure to sedative-hypnotic drugs
- Zopiclone: Exposure to sedative-hypnotic drugs; Patients who have taken Zopiclone for at least one week before the first date of enrollment
  Interventions: Drug: Exposure to sedative-hypnotic drugs
- Control Group: Patients not taking any of the included or any other anxiety-hypnotic agents

INTERVENTIONS:
Drug: Exposure to sedative-hypnotic drugs — These patients will have been prescribed a sedative-hypnotic drug for at least one week prior to enrollment.
  Other Names: Medication Exposure
  Groups: Alprazolam; Diazepam; Estazolam; Flunitrazepam; Lorazepam; Zolpidem; Zopiclone

SUMMARY:
The aims of this study are to (1) examine the medication use patterns of commonly prescribed hypnotics and the factors that were associated with the long-term and short-term use patterns among the elderly population in Taiwan; (2)investigate the associations of using hypnotics with the elderly patients' disease statuses, efficacy and safety, as well as its pharmacokinetic and pharmacogenetic characteristics;(3) determine the clinical, economic and humanistic outcomes of using hypnotics and the corresponding contributing factors for the elderly in Taiwan.

DETAILED DESCRIPTION:
Aging is associated with the changes in the sleep structure, continuity, and timing while it also affects the elderly's physiological and psychological health statuses. Despite the fact that hypnotics are beneficial for the short-term management of insomnia, it is inconclusive about the risk and benefit ratios of long-term use for the elderly. The objectives of this study are to (1)examine the medication use patterns of prescribed hypnotics and the factors that were associated with the use patterns among the elderly population; (2)investigate the associations of using prescribed hypnotics with the elderly patients' disease statuses, efficacy and safety, as well as their pharmacokinetic and pharmacogenetic characteristics;(3)determine the clinical, economic and humanistic outcomes and corresponding factors of using hypnotics for long-term and short-term use in Taiwanese elderly.

This proposed study is the second part of a larger project that consists of two main phases across four years. The first part will include a retrospective database analysis to examine the medication use patterns for sleep disorders and corresponding outcomes using three data sets. Elderly patients aged 65 or older and who received hypnotics for insomnia will be selected from Taiwan's National Health Insurance Research Database, National Health Interview Survey and China Medical University Hospital (CMUH) in-house databases. Focus will be placed on benzodiazepines (BZD) and BZD-receptor specific non-BZD agents (Z-drugs), but Chinese traditional medication used for insomnia will also be examined.

This study is the second part of the larger project. The investigators will conduct a longitudinal, prospective, observational cohort study over a period of two years. The focus of this study is the use of hypnotic BZD and Z-drugs on elderly insomnia patients. The study cohorts include elderly patients, aged 65 years or older, who have received services in the outpatient departments of China Medical University Hospital, Taichung, Taiwan, and who have been prescribed with a selected BZD or Z-drug for insomnia for at least one week. A control group cohort will also be recruited. Each recruited patient will be monitored and evaluated periodically for at least one year. Economic, clinical, and humanistic outcomes, as well as adherence to the hypnotics will be assessed and monitored. Safety and tolerability will be assessed by occurrence of adverse drug reactions. Pharmacokinetic properties and genotyping patterns will be also be evaluated using snapshot blood sampling after the 6th month of enrollment in the study. The clinical and humanistic outcomes measures will include changes in insomnia status, functional status changes, depression status, as well as over-all well-being using EuroQol 5D. Economic evaluation will compare total insurance and out-of-pocket expenses at baseline and at 12 months follow up.

ELIGIBILITY:
* Inclusion criteria

  1. Patients who have received services in the outpatient departments in CMUH for at least six months persistently before the recruitment,
  2. who are diagnosed with any types of sleep disorders within the outpatient medical records, using ICD-9 codes to identify.
  3. who have been prescribed, for at least one week before the index date of observation, with one of the selected BZD or Z-drugs: estazolam, lorazepam, diazepam, alprazolam, flunitrazepam, zolpidem or zopiclone.
  4. who agree to participate in this observation study and have signed informed consent
* Exclusion criteria

  1. Those elderly patients who were diagnosed with cancers, seizures, specific psychiatric disorders (e.g., dementia, schizophrenia, panic disorder, alcohol withdrawal syndrome) and neurological disorders (e.g., Parkinson) in the baseline and during observation period

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Longitudinal prospective observational cohort study
  Elderly patients receiving regular outpatient services at China Medical University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in sleep quality at 12 months | after 12 months of enrollment
  Clinical outcome, measured by a Chinese version of the Pittsburgh Sleep Quality Index
Number of participants with an occurrence of associated ADR | after 12 months of enrollment
  Safety and tolerably, as measured by patients that experience falls, hip/limb fracture, cognitive impairment, etc. during the 12 months of enrollment

SECONDARY OUTCOMES:
Snapshot measurement of plasma drug and drug metabolite concentrations | after 6 months of enrollment
  Pharmacokinetic evaluation by determining the levels of drug and metabolite in the patients plasma after established use
Snapshot measurement of urine drug and metabolite concentrations | after 6 months of enrollment
  Pharmacokinetic evaluation by determining the levels of drug and metabolite in the patients plasma after established use -- and clearance after the sixth-month recruitments.
Calculation of drug clearance using snapshot plasma and urine concentrations | after 6 months of enrollment
  Pharmacokinetic evaluation by determining the patient's clearance of the drug after established use
Proportion of patients with CYP3A5 mutations | after 6 months of enrollment
  Pharmacogenetic evaluation and and genotyping of CYP3A5 enzyme for all enrolled patients with consent
Changes from baseline in sleep quality at 6 months | after 6 months of enrollment
  Clinical outcome, measured by a Chinese version of the Pittsburgh Sleep Quality Index
Changes from baseline in Barthel Index at 6 months | after 6 months of enrollment
  Clinical outcome, as a measure of independence, measured by Barthel Index
Changes from baseline in Barthel Index at 12 months | after 12 months of enrollment
  Clinical outcome, as a measure of independence, measured by Barthel Index
Changes from baseline in IADL at 6 months | after 6 months of enrollment
  Clinical outcome, as a measure of functional ability, measured by Instrumental Activities of Daily Living
Changes from baseline in IADL at 12 months | after 12 months of enrollment
  Clinical outcome, as a measure of functional ability, measured by Instrumental Activities of Daily Living
Changes from baseline in EQ-5D-5L & EQ-5D-VAS at 6 months | after 6 months of enrollment
  Changes in humanistic variables, as measured by the EuroQol 5D tool
Changes from baseline in EQ-5D-5L & EQ-5D-VAS at 12 months | after 12 months of enrollment
  Changes in humanistic variables, as measured by the EuroQol 5D tool
Changes from baseline in MMAS-8 after 6 months | after 6 months of enrollment
  Changes in medication adherence, as measured by the Morisky Medication Adherence
Changes from baseline in MMAS-8 after 12 months | after 12 months of enrollment
  Changes in medication adherence, as measured by the Morisky Medication Adherence
Change from baseline in economic healthcare costs using NHI and out-of-pocket expenses at 12months | At 12 months after enrollment
  NHI covered costs for inpatient and outpatient care taken from NHI data for the twelve months prior to enrollment, compared to the 12 months during enrollment. Added with patients' out of pocket expenses on health care.
Changes from baseline in insomnia at 6 months | After 6 months of enrollment
  Clinical outcome, measured by a Chinese version of the Athens Insomnia Scale
Changes from baseline in insomnia at 12 months | After 12 months of enrollment
  Clinical outcome, measured by a Chinese version of the Athens Insomnia Scale

CONTACTS AND LOCATIONS:
Overall Officials: Hsiang-Wen Lin, PhD, Principal Investigator — Pharmacist, Associate Professor
Locations (1):
- China Medical University Hospital, Taichung, Taiwan